CLINICAL TRIAL: NCT04625608
Title: A Randomised Controlled Trial Examining the Effect of Premedicant Oral Paracetamol on Gastric Residual Volume and pH in Children, in the Context of a 1-hour Clear Fluid Fast
Brief Title: Effect of Premedicant Oral Paracetamol on Gastric Volume and pH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 266252
Record Dates: First submitted 2020-07-29; First posted 2020-11-12 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Fasting
Keywords: general anaesthesia; children; paracetamol
MeSH Terms: conditions — Fasting | interventions — Acetaminophen; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard care (Other): Participants in this arm shall receive 3.6 ml/kg of water a minimum of 1 hour prior to the induction of general anaesthesia. This is standard practice in the 2 participating institutions.
  Interventions: Other: Standard care
- Paracetamol arm (Experimental): Participants in this arm shall receive 3 ml/kg of water plus 15 mg/kg of oral paracetamol suspension a minimum of 1 hour prior to the induction of general anaesthesia.
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Drug: Paracetamol — Standard care of 3 ml/kg water, plus 15 mg/kg oral paracetamol suspension, a minimum of 1 hour prior to the induction of general anaesthesia.
  Arms: Paracetamol arm
Other: Standard care — Standard care of 3.6 ml/kg water, a minimum of 1 hour prior to the induction of general anaesthesia.
  Arms: Standard care

SUMMARY:
Patients are asked to fast before general anaesthesia to reduce the risk that any gastric contents could be regurgitated and aspirated into the lungs once anaesthetised. If aspiration does occur, the volume and acidity of the fluid aspirated are thought to determine the extent of any harm caused. Recent guidelines have reduced the required fasting time for children for clear fluids from 2 hours to 1 hour before induction of anaesthesia, as it is understood that this does not adversely affect the gastric residual volume or increase its acidity. Paracetamol is commonly used to relieve pain during and after surgery. Paracetamol syrup preparations used in children are viscous and not classified as clear fluid. This study seeks to establish whether there is non-inferiority in gastric residual volume (GRV) and pH in children receiving oral paracetamol one hour before induction of anaesthesia and those who do not, when both groups have received a set volume of diluted orange cordial to drink. It is anticipated that if shown to have little or no impact on GRV and pH, oral paracetamol syrup can be given to children before surgery. This will omit the need for IV paracetamol to be given in theatre, potentially reducing cost and the risk of drug errors.

DETAILED DESCRIPTION:
Patients are asked to fast before anaesthesia to reduce the risk that residual gastric contents could be regurgitated and aspirated into the lungs once anaesthetised. In animal studies, gastric contents that are less acidic (with a pH >1.8) have been shown to be less harmful when aspirated than those that are more acidic, even at higher gastric residual volumes. Recent European and UK guidelines have reduced the length of the recommended clear fluid fast to 1 hour for children, as there is no significant difference in GRV or pH in children fasted for 1 hour compared to 2 hours. It is therefore believed to present no additional risk of harm.

Some anaesthetists administer oral paracetamol syrup to children pre-operatively as an alternative to intravenous administration of paracetamol during their surgery. The oral route has been suggested to be pleasant for children, cheaper, more convenient, and reduce the risk of drug errors associated with the IV preparation. Anderson et al found no significant difference in gastric volume or pH in children with a mean age of 8.5 years given paracetamol orally 90 minutes before surgery compared to children given paracetamol rectally. Burke et al. demonstrated that giving paracetamol orally up to 8 minutes before induction of anaesthesia was not associated with an increase in the volume of stomach contents, and that the pH of stomach contents was higher than in control subjects who did not receive paracetamol. This suggests that giving oral paracetamol before induction of anaesthesia may not present any increased risk of harm from aspiration. This was in the context of a mean fluid fast of 5 hours and a mean age of 5.1 years.

To our knowledge, no studies have assessed the effect of oral paracetamol syrup on gastric residual volume (GRV) and pH in the context of the newly recommended reduced clear fluid fasting time of 1 hour. Neither has this been studied in children as young as 44 weeks post-conceptual age.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* Requiring tracheal intubation for general anaesthesia
* Parent/guardian able to speak and understand written English

Exclusion Criteria:

* Known or suspected gastro-intestinal disease including varices
* Previous surgery which may alter gastric emptying or the anatomy of the oesophagus or stomach
* Anticipated difficult airway
* Concomitant administration of any other medication orally prior to anaesthesia, but excluding buccal sedative pre-medication eg midazolam
* Bleeding disorders
* Patients taking antacids or pro-kinetic drugs, or requiring them pre-operatively
* Allergy to paracetamol
* Patient weight greater than 25 kg
* Parental or patient refusal

Ages: 44 Weeks to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 104 (Estimated)
Dates: Start 2020-10-06 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Residual volume of gastric contents following induction of general anaesthesia | Approximately 5-10 minutes following the induction of general anaesthesia.
  Gastric volume and pH of that fluid that can be aspirated via an oro-gastric tube, passed into the patient's stomach once general anaesthesia has been induced and the airway secured.
pH of gastric contents following induction of general anaesthesia | Approximately 5-10 minutes following the induction of general anaesthesia.
  Gastric volume and pH of that fluid that can be aspirated via an oro-gastric tube, passed into the patient's stomach once general anaesthesia has been induced and the airway secured.

OTHER OUTCOMES:
Adverse events at induction of anaesthesia | Up to 10 minutes after the induction of anaesthesia
  Adverse events occurring around the time of induction of anaesthesia including regurgitation and aspiration of gastric contents
Adverse events at emergence from anaesthesia | Up to 10 minutes from removal of the patient's airway
  Adverse events occurring around the time of emergence from anaesthesia including regurgitation and aspiration of gastric contents
Paracetamol drug errors | For day case patients, until discharge. For inpatients, up to 24 hours post-operatively.
  Paracetamol related drug errors
Emergence delirium | Up to 10 minutes following patient arrival in PACU.
  Incidence of emergence delirium in post-anaesthesia care unit, measured with PAED score.
Adverse events in Post-Anaesthesia Care Unit | From arrival in the post-anaesthesia care unit until patient is ready for discharge to the ward, up to 24 hours.
  Adverse regurgitation or aspiration events occurring in the post-anaesthesia care unit, including requirements for additional analgesia, time to first analgesic request and time spent in the post-anaesthesia care unit.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Saffer, MB BS, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thomas M, Morrison C, Newton R, Schindler E. Consensus statement on clear fluids fasting for elective pediatric general anesthesia. Paediatr Anaesth. 2018 May;28(5):411-414. doi: 10.1111/pan.13370. Epub 2018 Apr 27. PMID 29700894
- [Background] Brady M, Kinn S, O'Rourke K, Randhawa N, Stuart P. Preoperative fasting for preventing perioperative complications in children. Cochrane Database Syst Rev. 2005 Apr 18;(2):CD005285. doi: 10.1002/14651858.CD005285. PMID 15846750
- [Background] James CF, Modell JH, Gibbs CP, Kuck EJ, Ruiz BC. Pulmonary aspiration--effects of volume and pH in the rat. Anesth Analg. 1984 Jul;63(7):665-8. PMID 6731893
- [Background] Jibril F, Sharaby S, Mohamed A, Wilby KJ. Intravenous versus Oral Acetaminophen for Pain: Systematic Review of Current Evidence to Support Clinical Decision-Making. Can J Hosp Pharm. 2015 May-Jun;68(3):238-47. doi: 10.4212/cjhp.v68i3.1458. PMID 26157186
- [Background] Anderson BJ, Rees SG, Liley A, Stewart AW, Wardill MJ. Effect of preoperative paracetamol on gastric volumes and pH in children. Paediatr Anaesth. 1999;9(3):203-7. doi: 10.1046/j.1460-9592.1999.00348.x. PMID 10320598
- [Background] Burke CN, D'Agostino R, Tait AR, Malviya S, Voepel-Lewis T. Effect of Preemptive Acetaminophen Administered Within 1 Hour of General Anesthesia on Gastric Residual Volume and pH in Children. J Perianesth Nurs. 2019 Apr;34(2):297-302. doi: 10.1016/j.jopan.2018.05.015. Epub 2018 Sep 27. PMID 30270047
- [Derived] Saffer E, Nielsen DPD, Warwick E, Stilwell A, Webb C, Chow G, Place MK. Effect of pre-operative oral paracetamol on gastric residual volume and pH in young children in the context of a 1-hour clear fluid fast: a randomised controlled trial. Anaesthesia. 2022 Apr;77(4):449-455. doi: 10.1111/anae.15670. Epub 2022 Feb 15. PMID 35166373